CLINICAL TRIAL: NCT03226496
Title: A Pilot Study Assessing a Single Motivational Interviewing Session to Improve Uptake of PrEP Among Young Black Men Who Have Sex With Men
Brief Title: Motivational Interviewing for PrEP Uptake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Richard Crosby (Other)
Collaborators: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor-Investigator, Richard Crosby, Sponsor PI, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: #2015-0210
Record Dates: First submitted 2017-07-20; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: the Intervention Condition is a Brief Motivational Interviewing Session
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): This group receives a brief motivational interviewing session about PrEP
  Interventions: Behavioral: motivational interviewing
- Control Group (No Intervention): This group receives standard of care clinic based counseling about PrEP

INTERVENTIONS:
Behavioral: motivational interviewing
  Arms: Intervention Group

SUMMARY:
The aim of the proposed supplemental study is to test a single session motivational interviewing (MI) program designed to promote the acceptance and use of PrEP for high-risk young Black men who have sex with men (YBMSM) and to determine whether previous assignment to study condition moderates these outcomes.

DETAILED DESCRIPTION:
The aim of the proposed supplemental study is to test a single session motivational interviewing (MI) program designed to promote the acceptance and use of PrEP for high-risk young Black men who have sex with men (YBMSM) and to determine whether previous assignment to study condition moderates these outcomes. In the parent study we had the foresight to include a cross-sectional survey of men's attitudes toward PrEP use as part of their first follow-up assessment. Using that data, we will identify the predictors of readiness to accept PrEP and we will use these findings to inform the design of a brief Motivational Interviewing session (MI-PrEP) that will promote uptake of PrEP. We will enroll 65 YBMSM who have completed the 12-month follow-up assessment from the parent study and 35 YBMSM (same inclusion criteria) from either of two clinics used in the parent study (the Crossroads Clinic or the Open Arms Clinic) who did not participate in the parent study. Using small block randomization, these 100 men will be assigned to the MI-PrEP condition or to the standard of care only control condition. At the conclusion of the enrollment session men will be asked if they would like to schedule an appointment to begin taking PrEP. This same offer will be made again approximately 14 days after the enrollment session. The dependent variables will thus include measures of whether men made/kept an appointment to begin PrEP and, if so, how much time elapsed before doing so and whether they filled the prescription for PrEP. For those who do fill the prescription we will test their blood for levels of tenofovir and emtricitabine after 3 months of time has elapsed. Group differences (Intervention vs. Control) in uptake, time to uptake, and actual use/adherence of PrEP are hypothesized to favor those receiving the MI-PrEP intervention program. If this is the case then an initial body of evidence will exist supporting the potential efficacy of a Motivational Interviewing-based, single session intervention that can be delivered to YBMSM in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

self-identify as being Black/African American and they must be 18 to 29 years of age. In addition, these men must answer yes to the following screening question: "have you had anal sex with a male in the past 6 months?" Also, to be eligible all men (including those having completed the 12-month follow-up assessment in the parent study) must have an HIV-negative test result in the past 30 days.

Exclusion Criteria:

already taking PrEP

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01-03 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Obtains first prescription for PrEP | 3 months
  first prescription will be determined by self report